CLINICAL TRIAL: NCT05352464
Title: Effects of Cervical Traction With and Without EMG Biofeedback in Patients With Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC -01052 Sana Sabir
Record Dates: First submitted 2022-04-25; First posted 2022-04-28 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Cervical Radiculopathy
Keywords: cervical traction; Range of motion; pain; EMG biofeedback; disability
MeSH Terms: conditions — Radiculopathy; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical traction with EMG biofeedback (Experimental): Continuous traction for 15-20 minutes in sitting position on average at an angle of 15-25 degrees of cervical flexion or in the most pain-free position.
  Ask the patient to assume sitting position on a comfortable chair. Place surface electrodes of EMG biofeedback at the level of C5-6 Para spinal muscles to pick up the activity of the muscles and convert it to vis-ual and auditory impulses produced from the device. Tell the patient to try to relax the tension of the neck muscles as much as he can by lowering the visual and auditory impulses from the device
  Interventions: Other: cervical traction with EMG biofeedback
- cervical traction and conventional physical therapy (Active Comparator): Continuous traction for 15-20 minutes in sitting position on average at an angle of 15-25 degrees of cervical flexion or in the most pain-free position.
  Interventions: Other: cervical traction and conventional physical therapy

INTERVENTIONS:
Other: cervical traction with EMG biofeedback — Continuous traction for 15-20 minutes in sitting position on average at an angle of 15-25 degrees of cervical flexion or in the most pain-free position.
  Ask the patient to assume sitting position on a comfortable chair. Place surface electrodes of EMG biofeedback at the level of C5-6 Para spinal muscles to pick up the activity of the muscles and convert it to vis-ual and auditory impulses produced from the device. Tell the patient to try to relax the tension of the neck muscles as much as he can by lowering the visual and auditory impulses from the device
  Arms: cervical traction with EMG biofeedback
Other: cervical traction and conventional physical therapy — Continuous traction for 15-20 minutes in sitting position on average at an angle of 15-25 degrees of cervical flexion or in the most pain-free position
  Arms: cervical traction and conventional physical therapy

SUMMARY:
Cervical radiculopathy is a neurological condition which is caused by underlying musculoskeletal disorders including herniated disc and degenerative changes in cervical spine that results in narrowing or stenosis of intervertebral foramen. This narrowing leads to compression of nerve root at the respective foramen. The compressed nerve root produces symptoms like numbness, tingling, pain and motor weakness in neck and upper extremity. These symptoms appear at the dermatome and myotome distribution of the affected nerve root. Mostly the cervical radiculopathy is present unilaterally but in severe cases it can appear bilaterally where bony spurs are found at various levels and nerve root in under compression on both sides.

DETAILED DESCRIPTION:
Cervical radiculopathy is a neurological condition which is caused by underlying musculoskeletal disorders including herniated disc and degenerative changes in cervical spine that results in narrowing or stenosis of intervertebral foramen. This narrowing leads to compression of nerve root at the respective foramen. The compressed nerve root produces symptoms like numbness, tingling, pain and motor weakness in neck and upper extremity. These symptoms appear at the dermatome and myotome distribution of the affected nerve root. Mostly the cervical radiculopathy is present unilaterally but in severe cases it can appear bilaterally where bony spurs are found at various levels and nerve root in under compression on both sides.

The annual incidence rate of cervical radiculopathy is reported to be 107.3 per 100,000 of men and 63.5 per 100,000 of women. So accordingly, the condition is more common in males than females.

Although no definitive treatment plan for cervical radiculopathy has been developed, there is a general consensus in the literature that using manual therapy techniques in conjunction with therapeutic exercise is effective in terms of increasing function and active range of motion (AROM). The focus will most likely be on reducing pain and disability. Recent researches have shown that exercise therapy has the highest beneficial outcomes.

Treatment options for rehabilitation plan includes: Education and advice, Manual Therapy - PAIVMs (Passive Accessory Intervertebral Movements) / PPIVMs (Passive Physiological Intervertebral Movements) / NAGs (Natural Apophyseal Glides) / SNAGs (Sustained Natural Apophyseal Glides),Exercise Therapy - AROM, stretching and strengthening and Postural re-education Cervical traction and electromyography (EMG) biofeedback have been administered by many physiotherapists and positive outcomes are revealed. Traction not only relives nerve root compression but also helps in managing acute pain instantly whereas EMG biofeedback is used to generate an electrical feedback signal in response to muscle activation and helps patients to learn a more effective way of using their weak muscles

ELIGIBILITY:
Inclusion Criteria:

* Symptoms duration was more than one month up to six months.
* Radiculopathy due to muscle spasm.
* Radiculopathy due to postero-lateral disc herniation.
* Pain radiating with numbness and tingling sensations to both arms, forearms and hands.

Exclusion Criteria:

* Patients diagnosed with thoracic outlet syndrome, diabetes mellitus, and/or carpel tunnel syndrome.
* Patients had severe sensory and/or motor manifestations.
* Patients had manifestations of central cervical disc herniation.
* Congenital conditions of the cervical spine.
* Patients with contraindications to mobilization techniques and those with dizziness due to vertebrobasilar insufficiency or vestibular dysfunctions.
* Cervical Fractures.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS): | for six weeks
  It is a subjective tool used to measure intensity of pain. It starts from 0 meaning "No pain" to 10 meaning "Worst pain". The reliability and validity of VAS measured by ICC is 0.97 and 0.941 respectively.Assesment to be done on baseline,2nd week,4th week and 6th week.
Neck Disability Index (NDI) | for six weeks
  It is also a subjective tool used to evaluate neck disability. It ranks from 0 meaning "No pain" to 5 meaning "Worst imaginable pain". The reliability and validity if NDI measured by Cronbach's alpha is 0.89 and 0.60-0.70 respectively. Assessment to be done at baseline,2nd week,4th week and 6th week.
EMG biofeedback | for six weeks
  It is an electric device use to generate electrical feedback signals from activation of muscles. The reliability and validity of EMG biofeedback is 0.815-0.979 (19) and 0.781-0.907 respectively.Assesment to be done at baseline,2nd week,4th week and 6th week.
Inclinometer. | for six weeks
  Inclinometers have dials or digital readouts that display the angle at which the inclinometer is situated relative to the line of gravity.
  Inclinometer measurements of cervical flexion, extension, lateral flexion, and rotation were found to be reliable for all three methods with ICCs ranging from 0.89 to 0.94.Assesment to be done at baseline,2nd week,4th week and 6th week.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No